CLINICAL TRIAL: NCT02618759
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Efficacy and Safety of DSXS in Patients With Mild to Moderate Plaque Psoriasis
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of DSXS in Patients With Mild to Moderate Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSXS 1505
Record Dates: First submitted 2015-11-01; First posted 2015-12-01 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DSXS1505 (Experimental): To evaluate the therapeutic efficacy and safety of DSXS topical spray, 0.15%.
  Interventions: Drug: DSXS; Drug: Placebo
- Placebo (Placebo Comparator): Eligible patients will be randomized in a 1:1 ratio to Test or Placebo product.
  Interventions: Drug: DSXS; Drug: Placebo

INTERVENTIONS:
Drug: DSXS — active treatment
  Other Names: Active
Drug: Placebo — placebo treatment
  Other Names: vehicle

SUMMARY:
The purpose of this study is to evaluate the therapeutic efficacy and safety of DSXS compared to a Placebo (vehicle) in patients with mild to moderate plaque psoriasis.

DETAILED DESCRIPTION:
To evaluate the therapeutic efficacy and safety of dsxs topical spray, 0.15% (Taro Pharmaceuticals, U.S.A., Inc.) compared to a Placebo (vehicle) spray (Taro Pharmaceuticals, U.S.A., Inc.) in patients with mild to moderate plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* male and non-pregnant females, 12 years of age or older, with a confirmed diagnosis of mild to moderate plaque psoriasis

Exclusion Criteria:

* patient is< 12 years old.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DSXS1505 | Placebo
Started | 60 | 59
Completed | 58 | 54
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other Reasons | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSXS1505 | Placebo | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (15.2) | 57.3 (14.3) | 55.4 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 33 | 36 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 28 | 57
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 56 | 54 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Baseline Total BSA [Mean (Standard Deviation); unit: meters squared] | 2.0 (0.3) | 2.0 (0.3) | 2.0 (0.3)
%BSA Affected with Psoriasis [Mean (Standard Deviation); unit: percent of BSA] | 7.2 (1.5) | 7.5 (1.7) | 7.3 (1.6)
Baseline Investigator's Global Assessment (IGA) Score [Count of Participants; unit: Participants] — IGA is an overall assessment of the severity of a patient's case of plaque psoriasis, rated 0 to 5 as detailed in Appendix C of the protocol. A higher value represents a more severe case of plaque psoriasis.
  Participants
    Clear | 0 | 0 | 0
    Minimal | 0 | 0 | 0
    Mild | 16 | 10 | 26
    Moderate | 44 | 49 | 93
    Severe | 0 | 0 | 0
Baseline Total Lesion Severity Score (TLSS) [Mean (Standard Deviation); unit: units on a scale] — TLSS is a lesion assessment to determine severity of a plaque psoriasis lesion based on a summation of scores Erythema, Scaling, and Plaque Elevation (each rated 0 to 5 in severity). This is detailed in Appendix B of the study protocol. The minimum value is 0, and the maximum value is 15. A higher value indicates a more severe plaque psoriasis lesion. To be considered for inclusion in the study, the Target Lesion must have a Plaque Elevation sub-scale score of at least 2.
  units on a scale | 8.4 (1.4) | 8.4 (1.5) | 8.4 (1.5)
Baseline Scaling Score [Count of Participants; unit: Participants]
  Clear | 0 | 0 | 0
  Almost Clear | 1 | 3 | 4
  Mild | 15 | 15 | 30
  Moderate | 40 | 35 | 75
  Severe | 4 | 6 | 10
  Very Severe | 0 | 0 | 0
Baseline Erythema Score [Count of Participants; unit: Participants]
  Clear | 0 | 0 | 0
  Almost Clear | 1 | 1 | 2
  Mild | 15 | 16 | 31
  Moderate | 40 | 37 | 77
  Severe | 4 | 5 | 9
  Very Severe | 0 | 0 | 0
Baseline Plaque Elevation [Count of Participants; unit: Participants]
  Clear | 0 | 0 | 0
  Almost Clear | 0 | 0 | 0
  Mild | 14 | 11 | 25
  Moderate | 43 | 43 | 86
  Severe | 3 | 5 | 8
  Very Severe | 0 | 0 | 0
Baseline Psoriasis Area Severity Index (PASI) Score [Mean (Standard Deviation); unit: units on a scale] — The PASI is a composite score based on the severity of three different clinical signs of psoriasis (Erythema, Induration, and Scaling, each rated 0 to 4 in severity) in four different areas of the body (Head/Neck, Upper Limbs, Trunk, and Lower Limbs) multiplied by the percent of that specific body area affected multiplied by a weighting factor. The scale is explained in detail in the study protocol Appendix D. The minimum score would be 0 and the Maximum Score would be 72. A higher value would represent a more severe case of psoriasis.
  units on a scale | 5.8 (2.5) | 6.2 (2.4) | 6.0 (2.5)
Target Lesion Size (area) [Mean (Standard Deviation); unit: centimeters squared] | 48.7 (55.1) | 36.7 (26.3) | 42.7 (43.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Each Treatment That Have Clinical Success Based on IGA at Day 28 ± 2
Description: The number of patients in each treatment group that have clinical success. Clinical Success is at least a 2-grade improvement from the baseline IGA score. The minimum IGA value is 0, and maximum value is 5. A higher number represents a more severe case of plaque psoriasis. Patients are required to have an IGA score of 2 or 3 at baseline, so all clinical success IGA scores will be either 0 or 1.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS1505 | Placebo
Number analyzed (Participants) | 60 | 59
Participants | 10 | 3
Statistical Analysis 1: Comparison: DSXS1505 vs Placebo; Test type: Superiority; p = 0.0745, Cochran-Mantel-Haenszel

2. Primary Outcome: Number of Patients in Each Treatment That Have Treatment Success Based on TLSS at Day 28 ± 2
Description: The number of patients in each treatment group that have Treatment Success for the Target Lesion based on the TLSS sub-scale scores. Treatment Success is defined as a score of 0 or 1 for each of the three signs and symptoms (erythema, scaling and plaque elevation) for the Target Lesion. Each score has a minimum value of 0 and maximum value of 5, where a higher value represents a more severe sign or symptom. To be considered for inclusion in the study, the Target Lesion must have a plaque elevation score of at least 2.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS1505 | Placebo
Number analyzed (Participants) | 60 | 59
Participants | 8 | 4
Statistical Analysis 1: Comparison: DSXS1505 vs Placebo; Test type: Superiority; p = 0.2310, Cochran-Mantel-Haenszel

3. Secondary Outcome: Number of Patients in Each Treatment That Have Clinical Success Based on IGA at Day 28 ± 2 (Patients With a Baseline IGA Score of 3)
Description: The number of patients in each treatment group that have clinical success. Clinical Success is defined as at least a 2-grade improvement from the baseline IGA score. This measure is limited to patients with a baseline IGA score of 3, so any IGA score of 0 or 1 at Day 28 ± 2 would be a treatment success.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS1505 | Placebo
Number analyzed (Participants) | 44 | 49
Participants | 8 | 3
Statistical Analysis 1: Comparison: DSXS1505 vs Placebo; Test type: Superiority; p = 0.1059, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Patients in Each Treatment That Have Treatment Success Based on TLSS at Day 28 ± 2 (Patients With a Baseline IGA Score of 3)
Description: The number of patients in each treatment group that have Treatment Success for the Target Lesion based on the TLSS sub-scale scores. Treatment Success is defined as a score of 0 or 1 for each of the three signs and symptoms (erythema, scaling and plaque elevation) for the Target Lesion. Each score has a minimum value of 0 and maximum value of 5, where a higher value represents a more severe sign or symptom. To be considered for inclusion in the study, the Target Lesion must have a plaque elevation score of at least 2. This measure is limited to patients with a baseline IGA score of 3.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS1505 | Placebo
Number analyzed (Participants) | 44 | 49
Participants | 4 | 3
Statistical Analysis 1: Comparison: DSXS1505 vs Placebo; Test type: Superiority; p = 0.6962, Cochran-Mantel-Haenszel

5. Secondary Outcome: Number of Patients in Each Treatment That Have Clinical Success Based on IGA at Day 28 ± 2 (Patients With a Baseline IGA Score of 2)
Description: The number of patients in each treatment group that have clinical success. Clinical Success is defined as at least a 2-grade improvement from the baseline IGA score. This measure is limited to patients with a baseline IGA score of 2, so only an IGA score of 0 at Day 28 ± 2 would be a treatment success.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS1505 | Placebo
Number analyzed (Participants) | 16 | 10
Participants | 2 | 0
Statistical Analysis 1: Comparison: DSXS1505 vs Placebo; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel

6. Secondary Outcome: Number of Patients in Each Treatment That Have Treatment Success Based on TLSS at Day 28 ± 2 (Patients With a Baseline IGA Score of 2)
Description: The number of patients in each treatment group that have Treatment Success for the Target Lesion based on the TLSS sub-scale scores. Treatment Success is defined as a score of 0 or 1 for each of the three signs and symptoms (erythema, scaling and plaque elevation) for the Target Lesion. Each score has a minimum value of 0 and maximum value of 5, where a higher value represents a more severe sign or symptom. To be considered for inclusion in the study, the Target Lesion must have a plaque elevation score of at least 2. This measure is limited to patients with a baseline IGA score of 2.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS1505 | Placebo
Number analyzed (Participants) | 16 | 10
Participants | 16 | 10
Statistical Analysis 1: Comparison: DSXS1505 vs Placebo; Test type: Superiority; p = 0.1044, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 1 year, 7 months
Arm/Group | DSXS1505 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 3/60 | 3/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSXS1505 (N=60) | Placebo (N=59)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Application site pain (General disorders) | 0 (0) | 1 (1)
Application site paraesthesia (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT02618759/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT02618759/SAP_001.pdf